CLINICAL TRIAL: NCT07349485
Title: A PAC Post-Market Clinical Study to Demonstrate Color Change in the WoundCue™ Kit When an Elevated Inhibitory Bacterial and/or Fungal Load is Present in a Wound
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ParaNano, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PRT-001; NSR (Other: ParaNano)
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Wound Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - MolecuLightDX™ or MolecuLight i:X™ imaging and PCR testing data taken prior to consent (Active Comparator): Subjects must have visible fluorescence when using MolecuLightDX™ or MolecuLight i:X™ imaging.
  • Arm #1's Screening Visit requires that the standard of care MolecuLightDX™ or MolecuLight i:X™ imaging and PCR testing data taken prior to consent be obtained and used in the Study, as authorized by the Informed Consent.
  Interventions: Diagnostic Test: HCy-hex™: a hemicyanine-based (HCy) lipase-responsive dye
- Arm 2 - MolecuLightDX™ or MolecuLight i:X™ imaging prior to application (Active Comparator): Arm #2's Visit #1 requires that the Clinical Site scans wound with MolecuLightDX™ or MolecuLight i:X™ imaging prior to application of the WoundCue™ Kit.
  Interventions: Diagnostic Test: HCy-hex™: a hemicyanine-based (HCy) lipase-responsive dye

INTERVENTIONS:
Diagnostic Test: HCy-hex™: a hemicyanine-based (HCy) lipase-responsive dye — HCy-hex™: a hemicyanine-based (HCy) lipase-responsive dye with a labile ester linkage, enzymatically cleavable by bacterial lipase released from clinically relevant strains of bacteria

SUMMARY:
The purpose of this research is to test if the investigational ParaNano WoundCue Kit can detect elevated inhibitory bacterial and/or fungal loads.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1:

Subjects will be considered qualified for enrollment if they meet the following criteria:

Subjects and/or Legally Authorized Representative (LAR) must voluntarily provide written Informed Consent, consisting of reading, signing, and dating the Informed Consent document after the Principal Investigator, sub-Principal Investigator, or other designated Study Staff member has explained the Study procedures, risks, and contact information.

Able and willing to comply with all Study requirements.

Subject can be Male or Female but must be over 21 years of age.

Subject is currently under the care of a Primary Care Physician.

Subject has an anticipated survival of greater than two months.

Subject has a moderate to high exudate wound that has visible fluorescence when using MolecuLightDX™ or MolecuLight i:X™ imaging.

Arm 2:

Subjects will be considered qualified for enrollment if they meet the following criteria:

Subjects and/or Legally Authorized Representative (LAR) must voluntarily provide written Informed Consent, consisting of reading, signing, and dating the Informed Consent document after the Principal Investigator, sub-Investigator, or other designated Study Staff member has explained the Study procedures, risks, and contact information.

Able and willing to comply with all Study requirements.

Subject can be Male or Female but must be over 21 years of age.

Subject is currently under the care of a Primary Care Physician.

Subject has an anticipated survival of greater than two months.

Subject has a moderate to high exudate wound.

*For this Study, moderate exudate is defined as a wound that may require a dressing change 2-3 times a week based on provider judgement. Heavy exudate is defined as a wound that may require a dressing change 4 or more times a week based on provider judgement.

Exclusion Criteria:

* Subject's target treatment area has a surface area larger than 5 cm2.

Known sensitivity or allergy to the Study Device or adhesives/adhesive-related products.

Current use of topical ointments, including over-the-counter products and prescription drugs, on or near the intended treatment area.

Current use or recent history (within the past 14 days) of antibiotics, either oral, systemic, or topical.

Undergoing therapy with another investigational agent that may affect the WoundCueTM Kit's performance within thirty (30) days of Study Visit 1 or planned participation overlapping with this Study.

Women who are pregnant, breastfeeding, or intend to become pregnant during the course of the Study.

Medical condition that, in the opinion of the Principal Investigator, would preclude safe Subject participation in the Study.

Adults who, in the judgment of the Investigator, lack the capacity to provide informed consent for themselves

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-11-20 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint: | 48 hours after screening
  80% correlation (1:1) in detection of elevated inhibitory bacterial and/or fungal load by WoundCue™ Kit and confirmed by laboratory testing.